CLINICAL TRIAL: NCT03566420
Title: Knowledge, Personal Views and Experiences of a Group of Dental Interns Toward Physical Child Abuse: A Cross Sectional Study
Brief Title: Knowledge, Personal Views and Experiences of a Group of Dental Interns Toward Physical Child Abuse
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Salma Ali Hassan, Dentist, Cairo University
Other Study IDs: CEBD-CU-2018-06-43
Record Dates: First submitted 2018-06-12; First posted 2018-06-25 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Child Abuse

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
Scientific background ( Statement of the problem) :

Child abuse is a worldwide problem facing millions of children annually regardless their socio-economic level and culture, it affects the child's physical, mental health, well-being and development through his life (WHO, 2002).

The World Health Organization stated that 23% of children worldwide were physically abused in 2014 (WHO, 2014). In Egypt, children face different types of abuse, the 2014 Demographic Health Survey (DHS) shows that 93% of children aged 1 to 14 years old have been exposed to violent disciplinary practices, including psychological aggression and/or physical punishment (UNICEF Egypt, 2014).

Exclusively dentists are in strategic position to detect signs of child abuse as 50-70% of reported physical child abuse cases include head and neck trauma and 25% of physical abuse injuries occur in or around the mouth. In addition, dentists can notice the characteristic properties of the family because they have a continued relationship with pediatric patients and their families (Shannon et al., 2016).

Rationale for carrying out this study As published data about Knowledge, personal views and experiences of dentists toward physical child abuse in Egypt is sparse. This study will be conducted to cover this point among a group of dental interns in Egypt and highlight their role in detecting and reporting physical child abuse cases.

Benefits to the practitioners

* Increase the awareness of pediatric dentists about child abuse and highlight their role in detecting and reporting physical abuse cases.
* Knowledge about physical signs of abuse and how to act with these cases will give the dentists confidence in reporting decision.
* Discovering the main causes of dentists' hesitation in reporting diagnosed physical child abuse.

Benefits to the patient and population

* As 50-70% of reported physical abuse cases occur in the head and neck area (Shannon et al., 2016), so the dentist may be the first person to detect the physical abuse toward a child and help in protecting him from repeated injuries by his reporting.
* Asking the parents and the children about the physical signs that the dentist suspects may make the parent fear from reporting and stop his act.

DETAILED DESCRIPTION:
Review of literature :

Databases and websites as PubMed, Google were searched for relevant literature in English until October 2017 with key words "Child abuse, Child maltreatment, Physical child abuse, Violence against children, Dentists, pediatric dentists" Sonbol et al., 2011 conducted a study to assess Knowledge, educational experiences and attitudes towards child abuse amongst Jordanian dentists, using structured self-administered questionnaire. The target population was all dentists registered in the Jordanian Dental Association Council (general dentists and specialists) , the respondents were 256, 34% of them said that they had formal training in recognizing and reporting child abuse, and 42% had continuing education training on the topic, 50% of the dentists suspected a case of child abuse in the past 5 years, but only 12% reported their suspicions. The main reasons for not reporting suspicions of abuse were fear from anger of parents (43%), uncertainty about diagnosis (41%) and uncertainty about referral procedures (41%). Those dentists who had formal training in dental school and post-qualiﬁcation courses in child abuse were signiﬁcantly more likely to report suspicions.

Sousa et al., 2011 conducted a study to assess the attitudes and perceptions of dentists regarding child abuse, and to investigate professional characteristics associated with the identification of suspected child abuse. A self-administered questionnaire was sent to the 276 dentists (general dentists and specialists) in Pelotas, Brazil with response rate 68%. Most dentists (85.7%) had never suspected child abuse cases. Among those who suspected, 76.0% didn't report the cases to authorities. No differences were observed between sexes, years of graduation, types of licenses, and the frequency at which children were treated.

Harsimran et al., 2015 conducted a cross-sectional survey to general dentists in Moradabad city in India to assess their knowledge and attitude regarding child abuse and to identify the barriers in reporting these cases using self-administered questionnaire sent by mail to 120 of them the response rate was 97%. Questions pertaining to knowledge of dentists showed that nearly 89.7% of them were able to distinguish between accidental injury and physical abuse. The rate of detecting cases of child abuse by respondents was (60%), Lack of knowledge about dentist's role in reporting child abuse accounted to 55% in the reasons for hesitancy to report.

Rodrigues et al., 2015 conducted a systematic review to assess the perception, knowledge and attitude of dentists towards the detection and management of domestic violence against children (DVAC) cases. A systematic search was performed in 6 databases: PubMed, ScienceDirect, LILACS, SciELO, GoogleScholar, and OpenGrey. No restriction of language, time, and publication status was considered. The search resulted in 1.024 articles, of which 18 fit the eligibility criteria. The knowledge for detecting cases of DVAC obtained during the under graduation course was classified by the dentists (in 39% of the articles) as "insufficient". When suspecting of cases involving domestic violence, most of the dentists (in 77.75% of the articles) considered reporting to the competent authorities. However, the dentists were not sure about who these authorities are (in 31.25% of the articles).

Mogaddam et al., 2016 conducted a study to assess Knowledge, attitudes and behaviors of dentists regarding physical child abuse in Jeddah, Saudi Arabia, the target populations for this study were pediatric dentists, pediatric dentistry residents, and dental interns practicing in all of the dental schools in Jeddah. 270 self-administered questionnaires were distributed; the response rate was 77%. The participants showed insufficient knowledge of the signs and symptoms of child physical abuse, actions that should be taken in suspected cases, circumstances in which to report such cases, and the legal authorities to which they should be reported. The attitudes of participants towards detecting and reporting cases were generally positive. Only 11% of the participants had suspected a case of child abuse, and only 3% of them reported it. The main causes of under-reporting were lack of knowledge about referral procedures and fear of anger from family members.

Aim of the study :

The aim of this study is to:

Assess knowledge, personal views and experiences of a group of dental interns toward physical child abuse.

PO:

(P) Population: Dental interns that completed their Pediatric Dentistry round in Pediatric Dentistry and Dental Public Health Department , Faculty of Dentistry, Cairo University.

(O) Outcomes: Knowledge, personal views, experiences of dental interns toward physical child abuse.

Research question :

What is the knowledge, personal views and experiences of a group of dental interns toward physical child abuse

Study design: Cross-sectional study.

Study settings:

* Questionnaires, Appendix 1 will be distributed to the dental interns and give them 30 minutes to answer it.
* All questionnaires will be collected at the same day, to prevent any of the participants to search for the answers of questions that related to their knowledge.
* Participants during answering the questionnaire are not allowed to ask their colleagues, to ensure accuracy of the answers of knowledge questions.
* The researcher is not allowed to help the participant in answering the questions.
* Participants are allowed to ask the researcher any question either to clarify any part of the questions or anything about the survey.
* The researcher will deal with the participant personally, so there is no risk of the same dentist to complete more than one questionnaire.
* After the participants finish answering the questionnaires, it will be collected and subjected to statistical analysis.
* Data will be collected during 6 months.

Study size:

We are going to apply a convenient consecutive sampling; it will include all Dental interns at Faculty of Dentistry, Cairo University. Dental interns will be invited to complete the questionnaire. All number of interns will be reported, response rate will be calculated and no attempt is made to follow up with dental interns who were absent in the day of the survey.

Statistical methods:

Scores will be calculated according to the options selected by the intern dentists. The data will be analyzed using the statistical analysis software SPSS version 20. The individual scores will be summed up to yield a total score. Descriptive statistics will be calculated as mean scores, standard deviation and frequency distribution.

The difference of the oral health knowledge, attitude and practice between different categories will be assessed by Student's t-test or ANOVA according to the number of categories. The difference between male and female doctors will be assessed by student's t-test. P value < 0.05 will considered significant, All test will be 2 tails.

Ethical consideration

* A permission letter, explaining the aim of the study will be presented to the head of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University granting approval to conduct this survey .
* An informed consent explaining the aim of the study will be signed by the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Dental interns who completed their Pediatric Dentistry round in Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University.
2. Both genders are included.

Exclusion Criteria:

* Dental interns who refused to participate in the study.

Ages: 21 Years to 25 Years | Sex: All
Age Groups: Adult
Gender Based: Yes
Study Population: All dental interns that completed their Pediatric Dentistry round in Pediatric Dentistry and Dental Public Health Department , Faculty of Dentistry, Cairo University during 6 months period .
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2018-07 (Estimated); Primary Completion 2018-12 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Knowledge, personal views, experiences of dental interns toward physical child abuse | 6 months
  Measuring unit : Structured self-administered questionnaire (Sonbol et al., 2012, Dalledone et al., 2015 and Mogaddam et al., 2016)
  Measuring units : Numbers and percentages ( The questionnaire include binary and MCQ )

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Krug EG, Mercy JA, Dahlberg LL, Zwi AB. The world report on violence and health. Lancet. 2002 Oct 5;360(9339):1083-8. doi: 10.1016/S0140-6736(02)11133-0. PMID 12384003
- [Background] Mogaddam M, Kamal I, Merdad L, Alamoudi N. Knowledge, attitudes, and behaviors of dentists regarding child physical abuse in Jeddah, Saudi Arabia. Child Abuse Negl. 2016 Apr;54:43-56. doi: 10.1016/j.chiabu.2016.02.004. Epub 2016 Mar 15. PMID 26990176
- [Background] Owais AI, Qudeimat MA, Qodceih S. Dentists' involvement in identification and reporting of child physical abuse: Jordan as a case study. Int J Paediatr Dent. 2009 Jul;19(4):291-6. doi: 10.1111/j.1365-263X.2009.00971.x. Epub 2009 May 20. PMID 19476516
- [Background] Rodrigues JLSA, Lima APB, Nagata JY, Rigo L, Cericato GO, Franco A, Paranhos LR. Domestic violence against children detected and managed in the routine of dentistry - A systematic review. J Forensic Leg Med. 2016 Oct;43:34-41. doi: 10.1016/j.jflm.2016.07.006. Epub 2016 Jul 13. PMID 27441984
- [Background] Sonbol HN, Abu-Ghazaleh S, Rajab LD, Baqain ZH, Saman R, Al-Bitar ZB. Knowledge, educational experiences and attitudes towards child abuse amongst Jordanian dentists. Eur J Dent Educ. 2012 Feb;16(1):e158-65. doi: 10.1111/j.1600-0579.2011.00691.x. Epub 2011 May 5. PMID 22251340
- [Background] Azevedo MS, Goettems ML, Brito A, Possebon AP, Domingues J, Demarco FF, Torriani DD. Child maltreatment: a survey of dentists in southern Brazil. Braz Oral Res. 2012 Jan-Feb;26(1):5-11. doi: 10.1590/s1806-83242012000100002. PMID 22344331
- [Result] Kaur H, Vinod KS, Singh H, Arya L, Verma P, Singh B. Child maltreatment: Cross-sectional survey of general dentists. J Forensic Dent Sci. 2017 Jan-Apr;9(1):24-30. doi: 10.4103/jfo.jfds_6_15. PMID 28584471
- See also: Dalledone, M., de Paola, A.P.B., Correr, G.M., Pizzatto, E., de Souza, J.F. & Losso, E.M. (2015) Child abuse: Perception and knowledge by public health dentistry teams in Brazil. Brazilian Journal of Oral Sciences, 14 (3), pp.224-229. — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S1677-32252015000300224&lng=en&nrm=iso&tlng=en
- See also: Ajilian Abbasi, M., Saeidi, M., Khademi, G., Hoseini, B.L. & Emami Moghadam, Z. (2015) Child Maltreatment in the World: A Review Article. International Journal of Pediatrics, 3 (1.1), pp.353-365. — http://ijp.mums.ac.ir/article_3753_581.html